CLINICAL TRIAL: NCT02592070
Title: Activity & Cognition After Treatment (ACT) for Breast Cancer
Brief Title: Activity & Cognition After Treatment for Breast Cancer
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Edward McAuley, Shahid and Ann Carlson Khan Professor in Applied Health Sciences, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UIUC_IRB_15575
Record Dates: First submitted 2015-08-25; First posted 2015-10-30 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Mild Cognitive Impairment; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Motor Activity | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30 minute treadmill walking (Experimental): All participants will walk on the treadmill for 30 minutes and perform a battery of cognitive tasks immediately prior, immediately after, and one hour after completion of the 30 minute walking period.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — Participants will walk on the treadmill for 30 minutes at a moderate intensity.

SUMMARY:
This study addresses an important public health concern; impoverished cognitive function associated with treatment of breast cancer. Due to increased awareness of breast cancer combined with advances in medical care, there are over 2.8 million women living with a history of breast cancer in the U.S. alone. Chemotherapy and adjuvant therapy to remove cancerous tissue can result in deficits in attention, speed of processing, memory, and quality of life. Physical activity has been associated with a number of health benefits for breast cancer survivors including improvements in cognitive function. However, most of the literature is cross-sectional and it is unclear whether acute (single) bouts of physical activity affect cognition and, if they do, how long this effect lasts. This study will be the first, to the investigators' knowledge, to examine the effects of an acute bout of aerobic exercise on cognitive functioning in breast cancer survivors. Specifically, the investigators will determine the effects of a 30-minute moderate intensity aerobic exercise session (treadmill walking) on immediate and one hour follow up changes in measures of processing speed, memory, and executive function. Additionally, accelerometer cut-points for physical activity intensities in breast cancer survivors will be assessed. Finally, the investigators will examine the association of cardiorespiratory fitness and physical activity with changes in cognitive function. Findings from this study will allow researchers to determine whether any acute effects of exercise on cognition are retained over time and therefore have real meaning in the context of one's daily life.

DETAILED DESCRIPTION:
This study addresses an important public health concern: impoverished cognitive function associated with treatment of breast cancer. Due to increased awareness of breast cancer combined with advances in medical care, the 5-year survival rate has climbed to 89.2% with over 2.8 million women living with a history of breast cancer in the U.S. alone.

Unfortunately, the treatment of breast cancer is not without its consequences. Chemotherapy and adjuvant therapy to remove cancerous tissue can result in deficits in attention, speed of processing, memory, and quality of life. While past studies have identified memory and executive function as valuable, important determinants of long-term survival and quality of life in survivors of different types of cancer, it is unclear if standard care methods alone prove successful in attenuating declines in these variables. Previous research in breast cancer populations has found that executive function difficulties, namely in working memory, cognitive flexibility, and processing speed, as well as fatigue, are the most commonly described deficits. Furthermore, evidence suggests impairments in cognitive functioning may persist in up to 35% of breast cancer survivors years after treatment ends.

A behavioral and lifestyle modality known to improve physical and mental health status and protect against health declines is physical activity. Not only is physical activity known to protect against a host of diseases, but it also has been shown to provide many health benefits to breast cancer survivors. While the extant literature suggests that physical activity can lead to improvements in varying cognitive domains in breast cancer survivors, another study concluded that only 32% of these survivors meet the recommended guidelines for physical activity. Additionally, while benefits from physical activity for breast cancer survivors are well known, there is currently no scientifically recognized physical activity training program aimed at improving cognitive function in this cohort.

As such, a review chapter examining cognitive impairment in breast cancer survivors suggests more comprehensive studies examining the relationship between objective measures of physical activity, cardiorespiratory fitness, and cognitive performance are warranted to gain a better understanding of the potentially protective effects of fitness and physical activity on cognitive functioning in breast cancer survivors for better survival along the cancer continuum. In addition, other research has shown that subjective memory impairment, fatigue, and anxiety plague breast cancer survivors and suggests that breast cancer survivors may suffer from poorer quality of life as a result. Furthermore, it has been shown that breast cancer survivors have longer reaction time to working memory tasks compared to healthy, age-matched controls, and those survivors with higher levels of physical activity had shorter reaction times for more difficult tasks. A recent study also measured levels of objective physical activity and found those with higher levels displayed more positive measures of global cognition.

Despite this evidence, it is unknown if acute (single) bouts of exercise can provide benefits in varying cognitive domains. Previous research has shown that acute bouts of aerobic physical activity, of both light and moderate intensity, decrease state anxiety in breast cancer survivors. However, it is not known if these benefits extend to cognitive functioning. Furthermore, most of these results are founded in cross-sectional research and it is unclear whether acute bouts of physical activity improve cognition and, if they do, how long this effect lasts. This has implications for real world contexts in that, if benefits are present, breast cancer survivors can find relief in cognitive symptoms quickly by simply engaging in a bout of physical activity. This study will be the first, to the investigators' knowledge, to examine the effects of an acute bout of aerobic exercise on cognitive functioning in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* women between 30 and 60 years of age
* diagnosis of breast cancer
* no longer undergoing treatment
* fluent in English
* no history of dementia or organic brain syndrome
* not currently pregnant
* able to walk unassisted
* no health reasons that would prevent ability to exercise
* not currently enrolled in another exercise research study
* reported trouble with memory/concentration
* physician's consent

Exclusion Criteria:

* male
* no diagnosis of breast cancer
* outside of 30-60 years of age
* currently undergoing treatment for breast cancer
* inability to communicate in English
* history of dementia or organic brain syndrome
* pregnant
* unable to walk unassisted
* other health reasons that may prevent ability to exercise
* enrolled in another exercise research study
* no reported trouble with memory or concentration
* non-consent of physician

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cognitive function in breast cancer survivors immediately and one hour after an acute bout of exercise as assessed by a battery of cognitive functioning measures. | 1 year
  Participants will complete cognitive tasks, then exercise on a treadmill for 30 minutes before completing the same cognitive tasks again. Participants will then rest before completing the cognitive tasks one more time one hour after the end of the exercise period.

SECONDARY OUTCOMES:
Change in relationship between exercise and cognitive function in breast cancer survivors as assessed by physical activity and fitness levels. | 1 year
  The investigators wish to explore if participants with higher levels of fitness and higher levels of physical activity exhibit different levels of cognitive functioning compared to their less fit and less active peers.
Physical activity guidelines in breast cancer survivors as assessed by graded exercise test. | 60 minutes
  Participants will wear an accelerometer while performing a graded maximal exercise test. The output of the accelerometer will be compared to that of the exercise test to determine what levels of activity line up with varying metabolic equivalents. This will help us determine physical activity guidelines for breast cancer survivors.
Change from baseline in anxiety levels after one bout of exercise as assessed by HADS questionnaire. | 30 minutes
  Participants will complete a short anxiety questionnaire before and after a 30 minute bout of aerobic exercise. The investigators will then compare the pre- and post- values to examine if any changes are present.
Change in relationship between exercise and cognitive function in breast cancer survivors as assessed by psychosocial questionnaires. | 1 year
  Participants will take home a short battery of questionnaires designed to assess psychosocial outcomes. They will bring it back one week later. The investigators will then explore if participants with higher levels of any of these variables exhibit higher levels of cognition and/or fitness compared to peers with lower levels of psychological constructs.

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Freer Hall, University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, McCarron P, Parkin DM. The changing global patterns of female breast cancer incidence and mortality. Breast Cancer Res. 2004;6(6):229-39. doi: 10.1186/bcr932. Epub 2004 Aug 26. PMID 15535852
- [Background] Surveillance, Epidemiology, and End Results (SEER) Program (www.seer.cancer.gov) Research Data (2004-2010), National Cancer Institute, DCCPS, Surveillance Research Program, Surveillance Systems Branch, released April 2014, based on the November 2013 submission.
- [Background] van Harten WH, van Noort O, Warmerdam R, Hendricks H, Seidel E. Assessment of rehabilitation needs in cancer patients. Int J Rehabil Res. 1998 Sep;21(3):247-57. doi: 10.1097/00004356-199809000-00001. PMID 9812254
- [Background] Goodwin JS, Samet JM, Hunt WC. Determinants of survival in older cancer patients. J Natl Cancer Inst. 1996 Aug 7;88(15):1031-8. doi: 10.1093/jnci/88.15.1031. PMID 8683633
- [Background] Pinto AC, de Azambuja E. Improving quality of life after breast cancer: dealing with symptoms. Maturitas. 2011 Dec;70(4):343-8. doi: 10.1016/j.maturitas.2011.09.008. Epub 2011 Oct 19. PMID 22014722
- [Background] Kesler S, Hadi Hosseini SM, Heckler C, Janelsins M, Palesh O, Mustian K, Morrow G. Cognitive training for improving executive function in chemotherapy-treated breast cancer survivors. Clin Breast Cancer. 2013 Aug;13(4):299-306. doi: 10.1016/j.clbc.2013.02.004. Epub 2013 May 4. PMID 23647804
- [Background] Koppelmans V, Breteler MM, Boogerd W, Seynaeve C, Gundy C, Schagen SB. Neuropsychological performance in survivors of breast cancer more than 20 years after adjuvant chemotherapy. J Clin Oncol. 2012 Apr 1;30(10):1080-6. doi: 10.1200/JCO.2011.37.0189. Epub 2012 Feb 27. PMID 22370315
- [Background] Hillman CH, Erickson KI, Kramer AF. Be smart, exercise your heart: exercise effects on brain and cognition. Nat Rev Neurosci. 2008 Jan;9(1):58-65. doi: 10.1038/nrn2298. PMID 18094706
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Galantino ML, Greene L, Daniels L, Dooley B, Muscatello L, O'Donnell L. Longitudinal impact of yoga on chemotherapy-related cognitive impairment and quality of life in women with early stage breast cancer: a case series. Explore (NY). 2012 Mar-Apr;8(2):127-35. doi: 10.1016/j.explore.2011.12.001. PMID 22385567
- [Background] Baumann, F. T., Drosselmeyer, N., Leskaroski, A., Knicker, A., Krakowski-Roosen, H., Zopf, E. M., & Bloch, W. (2011). 12-week resistance training with breast cancer patients during chemotherapy: Effects on cognitive abilities. Breast Care, 6(2), 142-143.
- [Background] Irwin ML, McTiernan A, Bernstein L, Gilliland FD, Baumgartner R, Baumgartner K, Ballard-Barbash R. Physical activity levels among breast cancer survivors. Med Sci Sports Exerc. 2004 Sep;36(9):1484-91. PMID 15354027
- [Background] Mackenzie, M., Zuniga, K., & McAuley, E. (in press). Cognitive impairment in breast cancer survivors: The protective role of physical activity, cardiorespiratory fitness, and exercise training. Exercise-Cognition Interaction: Neuroscience Perspectives.
- [Background] Blacklock R, Rhodes R, Blanchard C, Gaul C. Effects of exercise intensity and self-efficacy on state anxiety with breast cancer survivors. Oncol Nurs Forum. 2010 Mar;37(2):206-12. doi: 10.1188/10.ONF.206-212. PMID 20189926
- [Derived] Salerno EA, Rowland K, Kramer AF, McAuley E. Acute aerobic exercise effects on cognitive function in breast cancer survivors: a randomized crossover trial. BMC Cancer. 2019 Apr 23;19(1):371. doi: 10.1186/s12885-019-5589-1. PMID 31014267
- See also: Exercise Psychology Laboratory website — http://www.epl.illinois.edu